CLINICAL TRIAL: NCT00734058
Title: Atrial Fibrillation Treatment Using Laser Ablation of Cardiac Tissue During Concomitant Cardiac Surgery
Brief Title: SOLAR & ATRILAZE Atrial Fibrillation Trial
Acronym: SAAF-T
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EndoPhotonix, Inc. (Industry)
Responsible Party: Kirk S Honour, Sr. Vice President, EndoPhotonix, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-AF-080808
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; AF; Atrial Fibrillation; Cardiac; Endocardial; Endocardium; EP; Electrophysiology; Epicardial; Epicardium; Heart; Interventional; Lesion; PVI; Pulmonary Vein; MAZE; Surgery; Surgical; Treatment; Patients with persistent AF with 3 months duration; Requiring concomitant open heart surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Persistent AF (Experimental): Treatment arm to be compared with historical control.
  Interventions: Device: Laser MAZE by Ablation of Cardiac Tissue

INTERVENTIONS:
Device: Laser MAZE by Ablation of Cardiac Tissue — The protocol calls for the creation of the pulmonary vein isolation lesion through the use of the SOLAR™. The additional lesions are to be created using the ATRILAZE™. At surgeon discretion, the ganglia may be ablated and left and right atrial appendages may be removed.
  Other Names: Maze; Maze procedure

SUMMARY:
The purpose of study is to conduct a pivotal evaluation of the EndoPhotonix™ SOLAR™ System and ATRILAZE™ System in order to obtain a labeling claim on the devices for the treatment of atrial fibrillation.

The study will test the safety and effectiveness of the EndoPhotonix™ Laser Ablation Systems to photocoagulate cardiac tissue during cardiac surgery, to create electrical isolation of the pulmonary veins and create other electrical isolation lesions in order to treat atrial fibrillation. The surgical procedure will be conducted during concomitant mitral valve repair or replacement surgery or in combination with other cardiac surgery including aortic valve surgery, tricuspid valve surgery, or coronary artery bypass surgery.

DETAILED DESCRIPTION:
The study objective is to generate Level II controlled data to support the expansion of indications for the SOLAR™ System based on 0-30 day data; as well as to support the expansion of indications for the SOLAR™ System and ATRILAZE™ System for the treatment of atrial fibrillation based on 180 days data. The data will be evaluated by comparing post-operative data to the historical control data. The subjects in the study cohort will receive laser ablation therapy using the investigational device during a concomitant surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Documented long term persistent atrial fibrillation (also known as permanent AF).of at least 3 months duration. Persistent AF is defined as AF which is sustained beyond seven days, or lasting less than seven days but necessitating pharmacologic or electrical cardioversion. Long term persistent AF is defined as continuous AF of greater than three months duration.
* Concomitant indication for open heart surgery for at least one of the following:

  * Mitral valve repair or replacement
  * Aortic valve repair or replacement
  * Tricuspid valve repair or replacement
  * Atrial septal defect (ASD) repair
  * Patent foramen ovale (PFO) closure
  * Coronary artery bypass procedure
* Be able to take anticoagulation therapy (Warfarin / Coumadin®)
* Be able to fulfill study requirements
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent

Exclusion Criteria:

* Life expectancy < 1 year
* NYHA class = IV
* Left ventricular ejection fraction (LVEF) measurement <30%
* Left atrial diameter > 7.5 cm
* Wolff-Parkinson-White (WPW) Syndrome
* Pregnancy or desire to be pregnant within 1 year of the study treatment
* Myocardial infarction within the previous 6 weeks
* Presence of a previously implanted device (valve, CS leads, or ICD)
* Known allergy, contraindication, or inability to comply with warfarin (Coumadin®) or heparin therapy
* Known allergy or contraindication to complying with anti-arrhythmic (Class IA, IC, III) therapy
* Previous thoracic procedure resulting in sternal opening and/or pericardial opening (e.g., CABG, valve replacement or repair)
* Current diagnosis of active endocarditis, local or systemic infection
* Renal failure requiring dialysis or hepatic failure
* Emergent cardiac surgery (cardiogenic shock)
* Preoperative need for intra-aortic balloon pump, IV inotropes or vasoactive agents
* Currently participating in another clinical research study
* Cerebral vascular accident or transient ischemic attack within previous 180 days or at any time with a documented residual neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation by 24-hour 3-lead Holter Monitor at the 180 day evaluation. On or Off Class 1 and III anti-arrhythmic medication | 180 days
Acute SAE: Death, mediastinitis, myocardial infarction, stroke, transient ischemic attack (TIA), pulmonary embolism, peripheral arterial embolism, esophageal injury, pulmonary vein stenosis; phrenic nerve damage | 0 through 30 days or length of stay

SECONDARY OUTCOMES:
SAE: Death, mediastinitis, myocardial infarction, stroke, transient ischemic attack (TIA), pulmonary embolism, peripheral arterial embolism, esophageal injury, pulmonary vein stenosis; phrenic nerve damage | 180 days
Determine binary freedom from AF, independent of anti-arrhythmic status as documented by 24 hour 3-Lead Holter Monitor. Reduction of AF burden with assumption of 100% initial burden. To establish improvement in Quality of Life. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Kirk S. Honour, Study Chair — EndoPhotonix, Inc.